CLINICAL TRIAL: NCT02838550
Title: Increasing Physical Activity Through a Motivational Online Intervention Using Pedometers in Sedentary Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rosa María Baños Rivera, Full Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H1466427733387
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Sedentary
Keywords: Physical Activity; Motivational Online Intervention; Pedometers
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- MOI and PEDOMETER (Experimental): Accessing to a motivational online intervention and wearing an unblinded pedometer (in order to receive feedback of the steps taken).
  Interventions: Behavioral: Motivational Online Intervention; Behavioral: Pedometer
- MOI (without PEDOMETER) (Experimental): Accessing to a motivational online intervention and wearing a blinded pedometer (in order to not receive feedback of the steps taken).
  Interventions: Behavioral: Motivational Online Intervention
- CONTROL (No Intervention): Wearing a blinded pedometer (in order to not receive feedback of the steps taken).

INTERVENTIONS:
Behavioral: Motivational Online Intervention — The self-administered Motivational Online Intervention developed by the authors was based on the "Transtheoretical Model of Change". It attempts to facilitate the decisional balance, the increase of the self-efficacy, and the use of experiential and behavioral processes of change (e.g., consciousness raising, counterconditioning, reinforcement management, stimulus control). The main objective is to deliver information to increase the motivation to practice physical activity and to set individualized goals. It has a total length of 45 minutes, and it is delivered in a web platform at the beginning of the intervention.
  Arms: MOI (without PEDOMETER); MOI and PEDOMETER
Behavioral: Pedometer — Wearing a pedometer of new generation that provides motivational messages from time to time to motivate the user to increase the physical activity, as well as information in the screen regarding all-day activity: steps taken, calories burned, distance travelled, floors climbed and active minutes.
  Arms: MOI and PEDOMETER

SUMMARY:
The aim of this study is to analyze the effect of a motivational online intervention (MOI) using pedometers to increase physical activity in a sample of sedentary students. It will be compared three conditions: MOI+PEDOMETER condition (access to a MOI and the use of a pedometer of new generation); MOI condition (access to a MOI and the use of a blinded pedometer); and CONTROL condition (the use of a blinded pedometer).

DETAILED DESCRIPTION:
Regular practice of physical activity (PA) has shown benefits in physical and mental health. However, the levels of PA are low in the general population. Pedometers and motivational online interventions (MOI) have been used to increase PA levels in sedentary population.

In spite of finding positive outcomes on PA levels when theoretical constructs derived from theories of behavior change and Internet have been used to guide pedometer-based interventions, few interventions have incorporated all these variables together and have analyzed the short-term or mid-term results.

The main objective of this study is to analyze the effect of a short self-administered Motivational Online Intervention (MOI) using pedometers to increase PA levels (primary outcome) and to change different theoretical constructs related to the PA behavior (positive decisional balance, self-efficacy, processes of change, stage of change, and enjoyment) (secondary outcomes) in a sample of sedentary students after 3-weeks intervention (post) and after 3-months (follow-up). It will be compared three conditions: MOI+PEDOMETER condition (access to a MOI and the use of a pedometer of new generation); MOI condition (access to a MOI and the use of blinded pedometer); and CONTROL condition (the use of a blinded pedometer). Hence, two conditions will include components of the "Transtheoretical Model of Change" in the intervention, such as the facilitation of the decisional balance, the increase of the self-efficacy, and the use of experiential and behavioral processes of change (e.g., consciousness raising, counterconditioning, reinforcement management, stimulus control), but only one of these condition will receive the feedback of the pedometer that will allow self-monitoring the behavior.

ELIGIBILITY:
Inclusion Criteria:

* to practice less than 30 minutes of moderate-intensity physical activity, three times a week;
* to be sedentary or low active (to walk less than 7500 daily steps during a week
* an age between 18 and 40 years old.

Exclusion Criteria:

* to be already using a pedometer;
* to suffer from a physical and/or a psychological disorder to prevent from practicing physical activity;
* to be already participating in other intervention to practice physical activity; and
* history of drug or alcohol addiction.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Daily Steps | Change from Baseline to Post-intervention (at 3 weeks) and Follow-up (at 3 months).

SECONDARY OUTCOMES:
Enjoyment of Physical Activity. Physical Activity Enjoyment Scale - Short Version (sPACES, Kendzierski & DeCarlo, 1991; Spanish adaptation of Fernández, Sánchez, & Bañuelos, 2008). | Change from Baseline to Post-intervention (at 3 weeks) and Follow-up (at 3 months).
Stages of change to practice Physical Activity. Stages of change questionnaire for exercise (SCQ; Marcus, Rossi, Selby, Niaura, & Abrams, 1992). | Change from Baseline to Post-intervention (at 3 weeks) and Follow-up (at 3 months).
Decisional balance to practice Physical Activity. Decision Balance Questionnaire for exercise (DBQ; Marcus, Rakowski, & Rossi, 1992). | Change from Baseline to Post-intervention (at 3 weeks) and Follow-up (at 3 months).
Self-efficacy to practice Physical Activity. Self-Efficacy Questionnaire (SEQ; Marcus, Selby, Niaura, & Rossi, 1992). | Change from Baseline to Post-intervention (at 3 weeks) and Follow-up (at 3 months).
Processes of change for Physical Activity. Processes of Change Questionnaire (PCQ; Marcus, Rossi, Selby, Niaura, & Abrams, 1992). | Change from Baseline to Post-intervention (at 3 weeks) and Follow-up (at 3 months).
Barriers to practice Physical Activity. Self-reported barriers to the practice of physical exercise (SBPPE, Niñerola, Capdevila, & Pintanel, 2006). | Baseline
Familiarity with the pedometers (ad-hoc questionnaire) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Baños, Full Prof., Principal Investigator — University of Valencia; Ausiàs Cebolla, PhD Ass., Study Chair — University of Valencia; Marta Miragall, PhD St., Study Chair — University of Valencia; Alejandro Domínguez, PhD St., Study Chair — University of Valencia; Jessica Navarro, PhD St., Study Chair — University of Valencia

IPD SHARING:
Plan to Share IPD: Undecided